CLINICAL TRIAL: NCT07264192
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of HS-10518 in Healthy Adult Premenopausal Females in China
Brief Title: A Study of HS-10518 in Healthy Adult Premenopausal Females in China
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: West China Second University Hospital (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Yu Qin, Director, Office of Clinical Trial Institution, West China Second University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HS-10518
Record Dates: First submitted 2025-11-16; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Infertility, Female
MeSH Terms: conditions — Infertility, Female

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- HS-10518 Dose 1 (Experimental): Dose level 1 of HS-10518, 10 mg Q12h, orally, 14 days
  Interventions: Drug: HS-10518
- HS-10518 Dose 2 (Experimental): Dose leve2 of HS-10518, 20 mg QD, orally, 14 days
  Interventions: Drug: HS-10518
- HS-10518 Dose 3 (Experimental): Dose leve3 of HS-10518, 20 mg Q12h, orally, 14 days
  Interventions: Drug: HS-10518
- HS-10518 Dose 4 (Experimental): Dose leve4 of HS-10518, 40 mg QD, orally, 14 days
  Interventions: Drug: HS-10518
- HS-10518 Dose 5 (Experimental): Dose leve5 of HS-10518, 80 mg QD, orally, 14 days
  Interventions: Drug: HS-10518
- Placebo (Placebo Comparator): placebo, BID, orally, 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HS-10518 — During the Dosing Period, four capsules of HS-10518 are administered twice daily at the same time points each day (morning and evening). The capsules should be swallowed whole with approximately 240 mL of water, and fluid intake is restricted within 1 hour before and after drug administration. Consecutive dosing should be maintained for 14 days.
  Arms: HS-10518 Dose 1; HS-10518 Dose 2; HS-10518 Dose 3; HS-10518 Dose 4; HS-10518 Dose 5
Drug: Placebo — During the Dosing Period, four capsules of HS-10518 Placebo are administered twice daily at the same time points each day (morning and evening). The capsules should be swallowed whole with approximately 240 mL of water, and fluid intake is restricted within 1 hour before and after drug administration. Consecutive dosing should be maintained for 14 days.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of HS-10518 in healthy adult premenopausal females in China

DETAILED DESCRIPTION:
In this randomized, double-blind, placebo-controlled Phase I clinical trial, 60 participants were randomized in a 1:1:1:1:1:1 ratio to receive HS-10518 (10 mg Q12h, 20 mg QD, 20 mg Q12h, 40 mg QD, or 80 mg QD) or placebo for 14 consecutive days. Assessments included safety, tolerability, PK parameters, and PD parameters.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be enrolled only if they meet all the following criteria:

  1. At the time of signing the informed consent form, the subject must be 18 to 40 years old (inclusive).
  2. Confirmed to be a healthy subject through medical assessment, including indicators such as medical history, physical examination, laboratory tests, and 12-lead electrocardiogram (ECG).
  3. Regular menstrual cycles for at least 6 months prior to screening, with:

     * Cycle length: 24 to 32 days;
     * Menstrual period duration: 2 to 7 days;(The first day of menstruation is defined as Day 1 of the menstrual cycle.)
  4. Baseline sex hormone levels meet the following requirements: Follicle-Stimulating Hormone (FSH) < 10 IU/L and Estradiol (E2) < 100 pg/mL; in addition, other sex hormone indicators must be assessed by the investigator as normal for the subject to be randomly enrolled.
  5. Body weight ≥ 45 kg, and Body Mass Index (BMI) within the range of 18 to 28 kg/m² (inclusive).
  6. The subject agrees to use highly effective non-hormonal contraceptive methods from the date of signing the informed consent form until 3 months after the administration of the last dose of the study drug. Highly effective non-hormonal contraceptive methods include:

     * Continuous abstinence;
     * Surgical sterilization of the subject (performed at least 3 months prior to signing the informed consent form);
     * Surgical sterilization of the subject's sexual partner (performed at least 6 months prior to signing the informed consent form).Other dual non-hormonal contraceptive methods are also acceptable, including:
     * Condoms with spermicides;
     * Diaphragms with spermicides (used with or without condoms);
     * Cervical caps with spermicides (used with or without condoms);
     * Vaginal sponges with spermicides (used together with condoms).
  7. Have a full understanding of the study content, process, and potential adverse reactions, and voluntarily sign the informed consent form.

Exclusion Criteria:

* Subjects will be excluded from the study if they meet any one of the following criteria:

  1. Has a history of abnormal uterine bleeding within 3 months prior to screening.
  2. Has never been sexually active.
  3. Has consumed foods or beverages rich in caffeine and/or xanthine (e.g., coffee, tea, chocolate, caffeinated carbonated beverages such as cola), tobacco-containing products (e.g., cigarettes), alcohol, or alcohol-containing products within 48 hours prior to drug administration.
  4. Has consumed grapefruit, grapefruit juice, bitter orange, bitter orange marmalade, bitter orange juice, or other products containing grapefruit or bitter orange within 7 days prior to the first dose.
  5. Has a history of smoking or alcohol abuse within 6 months prior to screening:

     * Smoking: More than 5 cigarettes per day or equivalent tobacco products;
     * Alcohol abuse: Alcohol consumption of ≥14 units per week (1 unit = 285 mL of beer, 25 mL of spirits with alcohol content ≥40%, or 150 mL of wine).
  6. Is suspected of substance abuse involving barbiturates, amphetamines, benzodiazepines, cocaine, opioids, cannabis, methadone, phencyclidine (PCP), tricyclic antidepressants (TCAs), or methamphetamine.
  7. Has a positive alcohol breath test or positive urine drug abuse screening result.
  8. Is pregnant, lactating, or has a positive serum beta-human chorionic gonadotropin (β-hCG) test at screening.
  9. Has a history of malignant tumors (cancer).
  10. Has had clinically significant gastrointestinal complaints, a history of gastrointestinal diseases (e.g., Crohn's disease, ulcerative colitis), or a history of surgery that may affect the absorption of the study drug (except for simple appendectomy or hernia repair) within 7 days prior to the first dose.
  11. Has a history of migraine, epilepsy, convulsions, depression, or a clinically significant depressive state.
  12. Has a history of thyroid or parathyroid dysfunction, or has thyroid-stimulating hormone (TSH), free triiodothyronine (FT3), or free thyroxine (FT4) levels outside the normal reference range-except if the investigator determines that the abnormality does not affect the study.
  13. Is within 6 months after childbirth, abortion, or cessation of lactation.
  14. Has a history of severe drug hypersensitivity, allergic diseases (e.g., asthma, urticaria, allergic rhinitis), or a history of atopy (allergic to ≥2 allergens)-if the investigator determines that the subject is unsuitable for the study.
  15. Has donated blood, lost ≥400 mL of blood, or received a blood transfusion within 3 months prior to screening; or has donated blood or lost ≥200 mL of blood within 1 month prior to screening.
  16. Has used any medications (prescription drugs, over-the-counter (OTC) drugs, traditional Chinese medicines, dietary supplements including vitamins, etc.) or short-term topical medications within 4 weeks prior to the first dose (or at least 5 times the respective elimination half-life, whichever is longer)-except if the investigator determines that the use does not affect the study.
  17. Has positive results for hepatitis B surface antigen (HBsAg), hepatitis C antibody (anti-HCV), human immunodeficiency virus antibody (anti-HIV), or syphilis serological test (TRUST)/treponema pallidum antibody (TP-Ab) at screening-except for subjects judged by the investigator to have a history of syphilis but have been cured.
  18. Has alanine transaminase (ALT) or aspartate transaminase (AST) levels exceeding the upper limit of normal (ULN) at screening.
  19. Has serum creatinine > 1.5 × ULN, or an estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m² (calculated using the Modification of Diet in Renal Disease (MDRD) formula) at screening.
  20. Has abnormal and clinically significant electrocardiogram (ECG) findings at screening (e.g., absolute value of QTcF [QT interval corrected by Fridericia's formula: QT/RR⁰·³³] > 470 milliseconds [ms]).
  21. Has diseases related to the ovaries, breasts, uterus, hypothalamus, or pituitary gland-if the investigator determines that the subject is unsuitable for the study.
  22. Has sonographic evidence of physiological abnormalities in the uterus and bilateral ovaries-if the investigator determines that the subject is unsuitable for the study.
  23. Has abnormal and clinically significant results from a cervical ThinPrep cytology test (TCT) during screening or within the past 12 months; for subjects with TCT results of "atypical squamous cells of undetermined significance (ASC-US)", enrollment is permitted only if high-risk human papillomavirus (HPV) testing is negative.
  24. Has recently used prohibited medications:

      * Used short-acting preparations containing sex hormones or affecting sex hormone levels (oral, transdermal, intravaginal, etc.) within 3 months prior to the first dose;
      * Used long-acting preparations containing sex hormones or affecting sex hormone levels (any long-acting injections or implants) within 6 months prior to the first dose.
  25. Plans to become pregnant during the study or within 3 months after the study ends.
  26. Participated in other clinical drug trials within 3 months prior to screening.
  27. Has other conditions or reasons deemed by the investigator to make the subject unsuitable for participation in the clinical study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2025-03-11 (Actual); Primary Completion 2025-06-23 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Area Under the Plasma Concentration-Time Curve from Time Zero to Time of Last Measurable Concentration (AUC0-t) of Metformin when administered alone | Days 1 to 4: From before the first dose to 30 hours after the last dose
  The AUC0-t of Metformin will be determined following multiple oral administrations of 0.5g Metformin twice daily for 3.5 days without XW003 coadministration.
Area Under the Plasma Concentration-Time Curve from Time Zero to Time of Last Measurable Concentration (AUC0-t) of Metformin when co-administered with XW003 at steady state | XW003 Steady-State Period ( Week 14): From pre-first dose of metformin to 30 hours post-last dose of metformin
  The AUC0-t of Metformin will be determined following multiple oral administrations of 0.5g Metformin twice daily for 3.5 days during the steady state of XW003 (1.2 mg weekly)
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-∞) of Warfarin when administered alone | D8: From pre-dose to 168 hours post-dose
  The AUC0-∞ of Warfarin will be determined following a single oral dose of 2.5 mg Warfarin without XW003 coadministration
rea Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-∞) of Warfarin when co-administered with XW003 at steady state | XW003 Steady-State Period (Week 16): From pre-dose of warfarin to 168 hours post-dose of warfarin
  The AUC0-∞ of Warfarin will be determined following a single oral dose of 2.5 mg Warfarin during the steady state of XW003 (1.2 mg weekly)

SECONDARY OUTCOMES:
Incidence of Adverse Events (AE) as assessed by CTCAE v5.0 | From screening to day 141
  The incidence, severity (graded by CTCAE v5.0), and relationship to the study drug of all adverse events (AEs), serious adverse events (SAEs), and AEs leading to study discontinuation will be recorded and summarized.
Number of Participants with Clinically Significant Changes in Laboratory Parameters | Baseline, Day 141
  Laboratory parameters include hematology, clinical chemistry, and urinalysis. The number and percentage of participants with clinically significant changes from baseline at each post-baseline visit will be summarized
Incidence of clinically significant abnormal findings in 12-lead electrocardiogram (ECG) | From screening to day 141
  Incidence of any clinically significant abnormal findings in 12-lead ECG is collected throughout study.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Qin, Principal Investigator — China West China Second University Hospital Chengdu, China
Locations (1):
- West China Second University Hospital, Chengdu, China